CLINICAL TRIAL: NCT00000905
Title: Discontinuation of Maintenance Therapy for Cytomegalovirus (CMV) Retinitis After Immune Reconstitution by Potent Antiretroviral Therapy: Safety, Virology, and Immunology Profiles
Brief Title: A Study to Evaluate the Effects of Stopping Maintenance Therapy for Cytomegalovirus (CMV) Retinitis After Effective Anti-HIV Therapy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 379
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2003-06

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Immunity, Cellular; Disease Progression; Cytomegalovirus Retinitis; DNA, Viral; Prognosis
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Disease Progression

SUMMARY:
The purpose of this study is to see if it is safe to stop maintenance therapy in HIV-positive patients with treated and healed CMV retinitis (eye disease) who have responded well to anti-HIV (antiretroviral) therapy.

The current therapies available to treat CMV retinitis are long-term therapies. However, it may be safe to stop long-term anti-CMV therapy in patients with healed CMV retinitis and stable CD4 counts resulting from taking a combination of at least 2 antiretroviral drugs.

DETAILED DESCRIPTION:
This study proposes to assess the hypothesis that, in HIV-infected patients with treated and healed CMV retinitis, an increase in CD4+ T-cells after initiation of potent antiretroviral therapy is either directly related to, or a marker of, immunologic protection for CMV retinitis and is associated with a recovery in specific proliferation responses to CMV antigens.

In this study, 100 patients [AS PER AMENDMENT 7/2/99: 50 patients] with treated and healed, non-immediate sight-threatening CMV retinitis will discontinue maintenance therapy for suppression of CMV retinitis. Patients are studied in 2 groups. Patients enrolled in Group 1 have CD4+ counts greater than 100 cells/mm3. Group 2 patients have CD4+ counts of 50-100 cells/mm3 and a minimum of a 2 log10 decrease in plasma HIV-1 RNA level or plasma HIV-1 RNA levels below the limit of detection while receiving potent antiretroviral therapy for at least 8 weeks prior to entry [AS PER AMENDMENT 7/2/99: Group 2 has been withdrawn]. An additional 25 patients who meet eligibility requirements but who choose to continue to receive maintenance therapy may also participate. All patients are followed to evaluate the relationship between reactivation or progression of CMV disease and changes in CMV DNA, HIV-1 RNA, and CD4+ cell counts. Patients are seen at Weeks 2, 4, 6 and 8, and every 4 weeks until study closure or for 12 months after the last subject is enrolled. [AS PER AMENDMENT 12/24/98: Patients with confirmed moderate to severe "immune recovery vitritis" should receive a 3-week course of systemic steroids (oral prednisone recommended). Moderate immune recovery vitritis is defined as symptomatic decrease in visual acuity of 2 or more Snellen lines along with, in the absence of active CMV disease, either 2+ or greater vitreous haze as defined by Nussenblatt et al., or cystoid macular edema.] [AS PER AMENDMENT 7/2/99: During the course of the study in patients with confirmed cystoid macular edema and a concomitant reduction in visual activity below 20/40, both attributable to immune recovery vitritis/uveitis only, a 21-day course of oral prednisone is recommended. This initial course of steroids helps to determine whether there is an improvement in vision or a decrease in macular edema. Long-term management of immune recovery vitritis/uveitis may include intraocular injection of steroids. Ophthalmoscopic examinations and laboratory tests are performed as per protocol.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 count greater than 100 cells/mm3.
* Have healed CMV retinitis after receiving anti-CMV therapy for at least 8 weeks within 3 months prior to study entry.
* Have taken antiretroviral therapy for at least 8 weeks prior to study entry; combination therapy must include at least 2 of the following: protease inhibitors (PIs), nucleoside reverse transcriptase inhibitors (NRTIs), or non-nucleoside reverse transcriptase inhibitors (NNRTIs).
* Have a life expectancy of at least 6 months.
* Are at least 13 years old (need consent if under 18).

Exclusion Criteria

You will not be eligible for this study if you:

* Have any unstable or severe medical conditions that would keep you from completing the study.
* Require chemotherapy or radiation therapy.
* Have a history of certain eye disorders.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75

CONTACTS AND LOCATIONS:
Overall Officials: Torriani F, Study Chair; Wohl D, Study Chair
Locations (25):
- United States (25):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Northwestern Univ Med School, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas Galveston, Galveston, Texas

REFERENCES:
- [Result] Wohl DA, Kendall MA, Owens S, Holland G, Nokta M, Spector SA, Schrier R, Fiscus S, Davis M, Jacobson MA, Currier JS, Squires K, Alston-Smith B, Andersen J, Freeman WR, Higgins M, Torriani FJ; ACTG 379 Study Team. The safety of discontinuation of maintenance therapy for cytomegalovirus (CMV) retinitis and incidence of immune recovery uveitis following potent antiretroviral therapy. HIV Clin Trials. 2005 May-Jun;6(3):136-46. doi: 10.1310/4J65-4YX1-4ET6-E5KR. PMID 16192248